CLINICAL TRIAL: NCT00299325
Title: A Randomized, Double Blind, Two-arm Placebo Controlled, 12-Month Study of the Effects of Rimonabant 20mg Once Daily on the Amount and the Activity of Visceral Fat in Abdominally Obese Patients With Metabolic Syndrome.
Brief Title: VIsceral Fat Reduction Assessed by CT-scan On RImonabAnt
Acronym: VICTORIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PM_C_0172; 2005-002568-27 (EudraCT Number)
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily with mild hypocaloric diet
  Interventions: Drug: Rimonabant; Other: Mild hypocaloric diet
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily with mild hypocaloric diet
  Interventions: Drug: Placebo (for Rimonabant); Other: Mild hypocaloric diet

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo
Other: Mild hypocaloric diet — Calculated by the dietitian based on the estimated basal metabolism rate and the physical activity

SUMMARY:
Primary objective:

To assess the effect of rimonabant on visceral fat area over a period of 12 months when prescribed with a mild hypocaloric diet in abdominally obese patients with metabolic syndrome

Secondary objectives:

* To assess the effect of rimonabant over a period of 12 months on:

  * Liver fat content using CT scan (Computed Tomography scan)
  * Anthropometric measures (weight, waist circumference, body composition using Dual Energy X-ray Absorptiometry (DEXA))
  * Lipid, lipoprotein profile
  * Glycemia, insulinemia and HbA1c
  * Adipokines, inflammatory and hemostatic markers
* To evaluate the percentage of patients with metabolic syndrome at 12 months
* To evaluate the safety and tolerability of rimonabant in these patients

In four selected US sites the effect of rimonabant at 12 months will be also assessed on:

* Basal lipolysis and insulin suppressed lipolysis (euglycemic hyperinsulinemic clamp).
* Resting metabolic rate and substrate oxidation at rest using indirect calorimetry.
* Adipose tissue histology and expression of genes involved in glucose and lipid metabolism (superficial adipose tissue biopsy).

DETAILED DESCRIPTION:
The total duration per patient will be approximately 15 months including a 12-month double-blind treatment period.

ELIGIBILITY:
Inclusion criteria :

* Waist circumference > 102 cm in men and > 88 cm in women
* Two other components of the metabolic syndrome (NCEP/ATPIII definition) among the following :

  * Triglyceridemia ≥ 150 mg/dl (or 1.69 mmol/L)
  * HDL cholesterol < 50 mg/dL (or 1.29 mmol/L) in women or < 40 mg/dL (or 1.04 mmol/L) in men
  * Blood pressure ≥ 130/85 mmHg (systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥ 85 mmHg) or Treatment with antihypertensive agent(s) for this condition
  * Fasting blood glucose > 110 mg/dl (or 6.1 mmol/L)

Exclusion criteria :

* Positive pregnancy test, pregnant or breast-feeding women, or women planning to become pregnant or breastfeed
* Absence of medically approved contraceptive methods for female of childbearing potential
* History of very low-calorie diet (≤ 800 kcal/day) within 3 months prior to screening visit
* History of surgical procedures for weight loss (eg, stomach stapling, bypass).
* Presence of any clinically significant endocrine disease according to the investigator.
* Weight change > 5 kg within 3 months prior to screening visit
* Obese patients (BMI> 40 kg/m²)
* Established type 1 or 2 diabetes (treated or untreated): at least 2 measures of fasting blood glucose ≥ 126 mg/dl
* Severe renal dysfunction (creatinine clearance < 30 ml/min) or nephrotic syndrome
* Chronic hepatitis or clinically significant hepatic disease
* Positive test for hepatitis B or C
* Marijuana or hashish users
* Significant haematology abnormalities (haemoglobin < 100 g/L and/or neutrophils < 1.5 G/L and/or platelets < 100 G/L).
* Presence or history of cancer within the past 5 years with the exception of adequately treated basal cell skin cancer or in situ uterine cervical cancer
* Presence or history of severe depression that can be defined as depression which necessitated the patient to be hospitalised, or patient with 2 or more recurrent episodes of depression or an history of suicide attempt
* Presence or history of bulimia or anorexia nervosa (DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria) or binge eating disorders
* Presence of any other condition (eg geographical, social…) current or anticipated that the Investigator feels that would restrict or limit the subject's participation for the duration of the studyRelated to previous or concomitant drugs that could interfere with the evaluation of study drug effects
* Administration of any investigational treatment (drug or device) within 30 days prior to screening
* Previous participation in a rimonabant study
* Administration of any of the following within 3 months prior to screening visit:

  * anti obesity drugs (eg, sibutramine, orlistat)
  * other drugs for weight reduction (phentermine, amphetamines)
  * herbal preparations for weight reduction
  * thyroid preparations or thyroxin treatment (except in patients on replacement therapy on a stable dose)
* Patient treated within the last 3 months with nicotinic acid, fibrates, bile acid sequestrants or ezetimibe (patients treated with statins can be included if the dose received is stable since at least 3 months and should not be modified during the whole study period).
* Patient treated with antidiabetic drug(s).
* Prolonged use (more than one week) within the last 3 months of systemic corticosteroids, neuroleptics, or antidepressants (including bupropion).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Relative change in visceral fat area assessed by CT scan | From baseline to Month 12

SECONDARY OUTCOMES:
Absolute change in visceral fat area assessed by CT scan | From baseline to Month 12
Change in Liver fat content measured using CT scan | From baseline to Month 12
Change in anthropometric measures | From baseline to Month 12
Change in specific lipid parameters | From baseline to Month 12
Change in glucose control parameters | From baseline to Month 12
Change in adipokines, inflammatory and hemostatic markers | From baseline to Month 12
Percentages of patients with a metabolic syndrome | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, MD, Study Director — Sanofi
Locations (9):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Hoersholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Stockholm, Sweden
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Result] Triay J, Mundi M, Klein S, Toledo FG, Smith SR, Abu-Lebdeh H, Jensen M. Does rimonabant independently affect free fatty acid and glucose metabolism? J Clin Endocrinol Metab. 2012 Mar;97(3):819-27. doi: 10.1210/jc.2011-2486. Epub 2011 Dec 14. PMID 22170727